CLINICAL TRIAL: NCT01823406
Title: Tissue-Specific Metabolic Reprogramming in Diabetic Complications. Glycemic Clamp Studies to Determine the Real Time Synthesis Rates of Glucose Derived Metabolites in Individuals With Type 1 Diabetes and Healthy Controls.
Brief Title: Tissue-Specific Metabolic Reprogramming in Diabetic Complications
Acronym: DP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Associate Professor Internal Medicine, MEND Division, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00060967; 1DP3DK094292-01 (NIH)
Record Dates: First submitted 2013-03-19; First posted 2013-04-04 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucose Clamp Technique; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Type 1 Diabetes no complications. (Experimental): Each cohort group will be admitted to the Michigan Clinical Research Unit for Blood glucose Clamp studies. Each subject will have a Euglycemic clamp (normal blood sugar clamp) for 4 hours and a hyperglycemic clamp (elevated blood sugar to 300) for 4 hours. Once the subject is clamped, bloods and urine will be collected to assay for specific metabolomics and proteomic biomarkers. We will perform the same clamps for each cohort.
  Interventions: Procedure: Euglycemic clamp (normal blood sugar clamp) for 4 hours; Procedure: hyperglycemic clamp (elevated blood sugar to 300) for 4 hours
- Type 1 Diabetes with microalbuminuria (Experimental): Each cohort group will be admitted to the Michigan Clinical Research Unit for Blood glucose Clamp studies. Each subject will have a Euglycemic clamp (normal blood sugar clamp) for 4 hours and a hyperglycemic clamp (elevated blood sugar to 300) for 4 hours. Once the subject is clamped, bloods and urine will be collected to assay for specific metabolomics and proteomic biomarkers. We will perform the same clamps for each cohort.
  Interventions: Procedure: Euglycemic clamp (normal blood sugar clamp) for 4 hours; Procedure: hyperglycemic clamp (elevated blood sugar to 300) for 4 hours
- Type 1 Diabetes with advanced complications. (Experimental): Each cohort group will be admitted to the Michigan Clinical Research Unit for Blood glucose Clamp studies. Each subject will have a Euglycemic clamp (normal blood sugar clamp) for 4 hours and a hyperglycemic clamp (elevated blood sugar to 300) for 4 hours. Once the subject is clamped, bloods and urine will be collected to assay for specific metabolomics and proteomic biomarkers. We will perform the same clamps for each cohort.
  Interventions: Procedure: Euglycemic clamp (normal blood sugar clamp) for 4 hours; Procedure: hyperglycemic clamp (elevated blood sugar to 300) for 4 hours
- Aged and sex matched healthy control volunteers (Experimental): Each cohort group will be admitted to the Michigan Clinical Research Unit for Blood glucose Clamp studies. Each subject will have a Euglycemic clamp (normal blood sugar clamp) for 4 hours and a hyperglycemic clamp (elevated blood sugar to 300) for 4 hours. Once the subject is clamped, bloods and urine will be collected to assay for specific metabolomics and proteomic biomarkers. We will perform the same clamps for each cohort.
  Interventions: Procedure: Euglycemic clamp (normal blood sugar clamp) for 4 hours; Procedure: hyperglycemic clamp (elevated blood sugar to 300) for 4 hours

INTERVENTIONS:
Procedure: Euglycemic clamp (normal blood sugar clamp) for 4 hours
Procedure: hyperglycemic clamp (elevated blood sugar to 300) for 4 hours

SUMMARY:
We will perform blood sugar studies to assess changes in metabolic (biochemical processes that occur within us) profiles associated with high blood sugar and diabetes.

DETAILED DESCRIPTION:
Objective: To assess steady state and dynamic metabolite changes in subjects with type 1 diabetes with and without microvascular complications and to understand intrinsic differences from non-diabetics in metabolite levels and flux.

The hypothesis is that diabetic complications arise from tissue-specific metabolic reprogramming resulting in alterations in fuel utilization which lead to dysfunction of the tissue. To test this hypothesis, we will use sensitive and specific mass spectrometer based metabolomic analysis to measure steady state metabolite levels in plasma and urine from controls subjects and subjects with T1DM, without and with diabetic complications during euglycemic and hyperglycemic clamp studies.

ELIGIBILITY:
Group 1: T1DM subjects without complications:

Group 2: T1DM subjects with microalbuminuria . Group 3: T1DM subjects with advanced diabetes complications Group 4: Age-and-sex-matched healthy control subjects .

Inclusion Criteria:

General entry criteria:

Must have type 1 diabetes > 5 years duration. 18 years of age or older

Subjects in the microalbuminuria group will have a history of urinary microalbumin to creatinine ration between 30-300 m/g confirmed on repeat testing while the non-albuminuric group will have a value of less than 30 mg/g.

Subjects in advanced complications group will have confirmed Retinopathy, Peripheral and/or Autonomic Neuropathy and nephropathy.

Non diabetic individuals will be matched for age and gender and will have normal glucose tolerance, normal lipid metabolism, and normal blood pressure.

Exclusion Criteria:

Age less than 18 . Women of child-bearing potential who may be pregnant or lactating History of pancreas, kidney or liver transplant History of drug or alcohol use. History of cancer other than basal cell carcinoma or squamous cell skin cancer. Presence of a condition that in the opinion of the investigator would make it unlikely for the subject to complete the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Difference in the levels of TCA cycle metabolites between groups during euglycemia and hyperglycemia | One time study visit /subject for an average of up to 24 h.
  Investigators will perform 4 hour Euglycemic and 4 hr hyperglycemic glucose clamps on each subject once. The Investigators will have 4 different groups of subjects. At specific time points during the clamps, the investigators will draw blood samples for measurement of metabolic assays and flux . The investigators will also collect spot urine samples for metabolic assay and flux.

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, MD,PhD., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States